CLINICAL TRIAL: NCT07078357
Title: Phase I/IIa Clinical Trial to Evaluate the Safety and Immunogenicity of StreptInCor, a Synthetic Vaccine Against Streptococcus Pyogenes, in Healthy Adult Volunteers.
Brief Title: Clinical Trial Phase I/IIa to Evaluate the Safety and Immunogenicity of StreptInCor
Acronym: StreptInCorVac
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Roney Orismar Sampaio, MD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 37164814.4.0000.0068
Record Dates: First submitted 2025-06-25; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Rheumatic Heart Disease; Rheumatic Heart Disease in Children; Vaccine Adverse Reaction; Rheumatic Diseases; Vaccine Acceptance; Vaccine
Keywords: Acute rheumatic fever; Rheumatic heart disease; Vaccine development program; Group A streptococcus (GAS); Streptococcus pyogenes
MeSH Terms: conditions — Rheumatic Heart Disease; Rheumatic Diseases; Rheumatic Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low dose Synthetic Vaccine Against Streptococcus Pyogenes- First arm (Experimental): 25 mcg / 50 mcg / 100 mcg / 200mcg of the experimental vaccine will be administered.
  Interventions: Other: Placebo
- Aluminum hydroxide (a vaccine adjuvant) - fifth arm (Placebo Comparator): Aluminum hydroxide (a vaccine adjuvant) will be administered as a placebo
  Interventions: Biological: StrepIncor; Other: Placebo

INTERVENTIONS:
Biological: StrepIncor — This arm will include 25/50/100/200 µg compared to placebo
  Arms: Aluminum hydroxide (a vaccine adjuvant) - fifth arm
Other: Placebo — A placebo (aluminum adjuvant) will be administered and compared to the other study arms

SUMMARY:
This is a Phase I/IIa, randomized, double-blind, placebo-controlled, dose-escalation clinical trial to test the candidate vaccine StreptInCor. The study will include four different doses (25 µg, 50 µg, 100 µg, and 200 µg) of StreptInCor produced under Good Manufacturing Practices (GMP) and formulated with aluminum hydroxide as the vaccine adjuvant. The adjuvant alone will be used as a placebo in this trial. Five groups, each consisting of twelve healthy adult volunteers, will randomly receive two doses of the vaccine or placebo with a 28-day interval, along with a booster dose six months after the initial vaccination

DETAILED DESCRIPTION:
This is a Phase I/IIa, randomized, double-blind, placebo-controlled, dose-escalation clinical trial to test the candidate vaccine StreptInCor. The study will include four different doses (25 µg, 50 µg, 100 µg, and 200 µg) of StreptInCor produced under Good Manufacturing Practices (GMP) and formulated with aluminum hydroxide as the vaccine adjuvant. The adjuvant alone will be used as a placebo in this trial.

Five groups, each comprising twelve healthy adult volunteers, will randomly receive two doses of the vaccine or placebo with a 28-day interval, along with a booster dose six months after the initial vaccination.

During the selection process, volunteers aged 18 to 45 years will undergo a general health assessment and serological tests to verify the absence of HIV and autoimmune diseases. Exclusion criteria include second-degree relatives or history of Rheumatic Fever (RF) or Rheumatic Heart Disease (RHD), as well as prior infections or recurrent diseases associated with S. pyogenes. All volunteers must sign an informed consent form before any procedures.

In the first phase of the trial, volunteers assigned to receive the lowest dose (25 µg) and three placebo volunteers will begin the vaccination scheme, maintaining blinding. One month after the second vaccination, all volunteers will be re-evaluated for safety, and the results will be submitted to the Data Safety Monitoring Committee (DSMC) for review. Only with a favorable opinion from the DSMC will the booster dose be administered to this group.

After the DSMC assesses the safety of these three doses, the second phase can commence. In this phase, volunteers assigned to the low-intermediate dose (50 µg) and three placebo volunteers will start vaccination, with safety evaluations occurring one month after the second dose. If the DSMC's opinion remains favorable, a booster at six months will be administered and re-evaluated by the DSMC.

If approved, the third phase will include the high-intermediate dose (100 µg) plus three placebo volunteers, with similar safety assessments and DSMC approval for the booster.

The fourth phase will involve volunteers receiving the high dose (200 µg) plus three placebo volunteers, following the same safety evaluation process.

In total, 60 volunteers will be enrolled - 12 per group and 15 per phase. Safety (toxicity) will be monitored by the DSMC after each booster at all protocol stages. The DSMC's operational procedures are based on the Ministry of Health's Guidelines for Data and Safety Monitoring Committees (2008). Safety parameters include serological markers for autoimmune diseases, with safety follow-up extending up to twelve months post-initial vaccination.

The study can be paused at any point if moderate or severe adverse events possibly related to the vaccine occur; in such cases, the DSMC will assess whether the trial or specific steps can be restarted.

The primary efficacy parameter will be at least a fourfold increase in IgG antibody levels after the last vaccination compared to pre-vaccination levels. All samples from the same volunteer will be assessed simultaneously to prevent processing bias, in a blinded manner. Additional efficacy measures include detection of other antibody classes, functionality of antibodies regarding surface binding and inhibition of bacterial invasion/adherence, induction of phagocytosis, cellular immune responses such as cytokine production, antigen-specific T-cell proliferation, and memory T-cell induction.

The dose showing the highest seroconversion rate and an acceptable rate of adverse effects will be selected for Phase II.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy male or female volunteers, aged between 18 and 45 years;

  * Availability to undergo all procedures throughout the study period;
  * Provide free and informed consent to participate in the study.

Exclusion Criteria:

* Participation in clinical trials within the last year
* Participation in cohort studies
* Diagnosis of concomitant infections or diseases that may affect immunity, including active HIV infection, hepatitis B, hepatitis C, diabetes mellitus, neoplasms, and autoimmune diseases;
* Current or previous diagnosis or family history of ARF, chorea, obsessive-compulsive disorder, or glomerulonephritis;
* Current or previous diagnosis of heart diseases;
* Severe asthma or chronic obstructive pulmonary disease (COPD);
* Abnormal neurological clinical assessment, especially chorea;
* Use of treatments that may affect immunity in the last four weeks, including immunomodulators, corticosteroids (only systemic use for two weeks or more), or antineoplastic agents;
* Use of treatments that may affect heart valves in the last four weeks or planned during the study period, including fenfluramine and dexfenfluramine;
* Renal insufficiency determined by estimated creatinine clearance below 45 ml/min/1.73m²;
* History of intolerance or allergy to any component of the study product, including antigen or adjuvant;
* Presence of valve abnormalities or alterations in cardiac anatomy as defined by echocardiogram;
* Altered electrocardiogram;
* Evidence or suspicion of recent S. pyogenes infection based on clinical symptoms in the last four weeks;
* Pregnancy, breastfeeding mother, or intention to become pregnant during the study period (only female participants);
* Any other condition that may interfere with the study process as assessed by the researchers, including sample size and statistical power.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | From enrollment to the end of treatment at six months
  • Safety outcome: The primary safety objective will be the absence of serious adverse events following immunization that have a reasonable causal relationship with the studied product in the StreptInCor and placebo groups;
Immunogenicity outcome | From enrollment to the end of treatment at six months
  Immunogenicity outcome: The primary immunogenicity outcome will be an increase of at least 4 times in IgG antibody levels against the StreptInCor peptide, 6 months after the last immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Kalil Filho, Full Professor, MD, PhD, Study Director — Heart Institute - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Heart Institute - Hospital Das Clinicas Da Faculdade de Medicina Da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We consider that, at this stage, individual participant data is confidential. However, these data may be made available in the future in accordance with the recommendations of our ethics committee

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT07078357/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT07078357/ICF_001.pdf